CLINICAL TRIAL: NCT02605681
Title: Plasma Midkine Associated Organ Dysfunction and Vascular Injury in Sepsis
Brief Title: Midkine and ACE-Ang II Induced Endothelial Injury in Sepsis
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Nanjing Zhongda hospital,Southeast University, China, Southeast University, China
Other Study IDs: 2015ZDSYLL069.0
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sepsis
Keywords: midkine; endothelial injury; sepsis; angiotensin-converting enzyme; angiotensin II
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- septic patients: We recruited the patients admitted to the Department of Critical Care Medicine, Zhongda Hospital, a tertiary hospital, from November 2017 to March 2018. The inclusive criteria were adult patients (age > 18 years-old and < 80 years-old) diagnosed with sepsis, according the definition of the Surviving Sepsis Campaign (2016). Exclusive criteria included: 1. age < 18 years-old or > 80 years-old; 2. pregnancy or breastfeeding; 3. malignancy; 4. patients with potentially elevated plasma midkine apart from sepsis including acute myocardial infarction, stroke, limb thrombosis, chronic renal dysfunction (baseline plasma creatine ≥2 mg/dL), autoimmune diseases and Alzheimer syndrome; 5. patients deceased or discharge from ICU within 24 hours; or, 6. written consents could not be obtained.

SUMMARY:
Plasma midkine has reported to be elevated in infection and a regulator of angiotensin-converting enzyme (ACE). We aimed to investigate the plasma midkine in septic patients and its association with 28-day mortality and organ function, and also with plasma ACE and angiotensin II.

DETAILED DESCRIPTION:
This study showed that Ang II induced endothelial injury in sepsis patients. Midkine has been shown to regulate the renin-angiotensin system and acts in the upstream signaling pathway of angiotensin (ANG) II. The investigators want to access the relationship between midkine level and ACE-Ang II induced endothelial injury in sepsis

ELIGIBILITY:
The inclusive criteria were adult patients (age > 18 years-old and < 80 years-old) diagnosed with sepsis, according the definition of the Surviving Sepsis Campaign (2016)

Exclusive criteria included: 1. age < 18 years-old or > 80 years-old; 2. pregnancy or breastfeeding; 3. malignancy; 4. patients with potentially elevated plasma midkine apart from sepsis including acute myocardial infarction, stroke, limb thrombosis, chronic renal dysfunction (baseline plasma creatine ≥2 mg/dL), autoimmune diseases and Alzheimer syndrome; 5. patients deceased or discharge from ICU within 24 hours; or, 6. written consents could not be obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed for sepsis
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
28-day mortality | up to 28 days
  All the patients were followed-up to 28 days and all-cause mortality was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu JY, Chang W, Sun Q, Peng F, Yang Y. Pulmonary midkine inhibition ameliorates sepsis induced lung injury. J Transl Med. 2021 Feb 27;19(1):91. doi: 10.1186/s12967-021-02755-z. PMID 33639987